CLINICAL TRIAL: NCT00103714
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, 28-Day Study of Denufosol Tetrasodium (INS37217) Inhalation Solution in Patients With Cystic Fibrosis Lung Disease
Brief Title: Study of Denufosol Tetrasodium in Patients With Cystic Fibrosis Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-104
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
Keywords: lung disease
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases | interventions — denufosol tetrasodium

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217)

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability and preliminary efficacy of two dose levels of INS37217 (denufosol tetrasodium) Inhalation Solution in patients with cystic fibrosis (CF) lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of CF
* Have an FEV1 greater than or equal to 60% or less than or equal to 90% of predicted normal
* Have oxygen saturation greater than or equal to 90% on room air
* Be clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation
* Be able to reproducibly perform spirometry maneuvers

Exclusion Criteria:

* Have changed their physiotherapy technique or schedule within 7 days prior to screening
* Have clinically significant comorbidities
* Using prior and concurrent medications according to the protocol

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2005-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
respiratory function

SECONDARY OUTCOMES:
adverse events
change in standard safety parameters
respiratory symptoms via questionnaire
pulmonary exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Amy Schaberg, BSN, Study Director